CLINICAL TRIAL: NCT01520792
Title: Paracétamol and Pharmacogenetic in Healthy Volunteers
Brief Title: Paracetamol and Pharmacogenetic
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0101
Record Dates: First submitted 2011-08-30; First posted 2012-01-30 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
Keywords: pharmacogenetic of paracetamol; Pain threshold
MeSH Terms: interventions — Acetaminophen; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paracetamol (Experimental)
  Interventions: Drug: Paracetamol (drug)

INTERVENTIONS:
Drug: Paracetamol (drug) — Randomized, single-center, placebo-controlled, double-blind, cross-over in 100 healthy volunteers meeting the inclusion criteria and receiving 2g of paracetamol orally or placebo on two study periods separated by one week.

SUMMARY:
Recent works has emphasized that the mechanism of action of paracetamol analgesic depend on its metabolism in the body, since a breakdown product of paracetamol, the AM404 is now considered the analgesic metabolite of paracetamol suggesting as paracetamol may be a pro-drug.

Indeed, it has been shown that paracetamol may have a deleterious effect, especially in vulnerable populations (hepatic insufficiency, elderly). First results showed a very significant decrease in sulfatation and gluthatione and increased phase 1 metabolism of acetaminophen, which involves enzymes such as cytochrome P450.

Multifactorial causes, combining nutrition (depletion of sulfur amino acids), increased detoxification of toxic metabolites of paracetamol, stress or trauma are discussed to explain the results.

Clinical studies showed a great variability of pain assessment by patients and variability in the metabolic response of paracetamol. Genetic factors probably play a role remains largely unknown.

The review of the literature on genetic polymorphism shows the involvement of a number of enzymes that are well known, predominantly on the metabolism of acetaminophen liver, but without connection with its analgesic effect. This is a critical missing link in the understanding of the analgesic effect of paracetamol.

DETAILED DESCRIPTION:
Randomized, single-center, placebo-controlled, double-blind, cross-over in 100 healthy volunteers meeting the inclusion criteria and receiving 2g of paracetamol orally or placebo on two study periods separated by one week.

The evaluation criterion is the difference in areas under the curve of pain thresholds to thermal and mechanical stimulations test

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Males
* Aged between 18 and 30 years

Exclusion Criteria:

* Subject without cons-indications of paracetamol

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Correlation between Pharmacogenetic profile and pain threshold | until 14 days before the administration

SECONDARY OUTCOMES:
Measures of thermal and mechanical pain thresholds | until 1 hour before the administration
Determination of blood concentration of gluthatione | until 1 hour before administration

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Pickering G, Creveaux I, Macian N, Pereira B. Paracetamol and Pain Modulation by TRPV1, UGT2B15, SULT1A1 Genotypes: A Randomized Clinical Trial in Healthy Volunteers. Pain Med. 2020 Apr 1;21(4):661-669. doi: 10.1093/pm/pnz037. PMID 30908574